CLINICAL TRIAL: NCT07324447
Title: CLINICAL TRIAL ON THE EFFECT OF SUPERVISED PHYSICAL EXERCISE AFTER BARIATRIC SURGERY ON MUSCLE MASS AND BONE DENSITY (OBEFIT STUDY)
Brief Title: EFFECTS OF SUPERVISED PHYSICAL EXERCISE AFTER BARIATRIC SURGERY ON MUSCLE MASS AND BONE DENSITY (OBEFIT STUDY)
Acronym: BARIATRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, Isaías Alarcón de Agua, Principal Investigator and Coordinator of the Esophagogastric and Bariatric Surgery Unit, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBEFIT STUDY
Record Dates: First submitted 2025-09-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Obesity &Amp;Amp; Overweight; Bariatric Surgery; Physical Exercise
Keywords: Obesity Surgery; Physical exercise; Bariatric Surgery
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical exercise program (Active Comparator): he primary objective is to try to minimise the loss of muscle mass that occurs in the patient. During the first 4 weeks of training, the objective is to familiarise the patient with the type of training to be carried out. The patient will do an initial block of strength work, followed by a block of cardiovascular work on a cycloergometer (continuous and variable) in the same session. Work will be done in order to progress in volume and intensity. Training sessions of approximately 50-60 minutes will be carried out 2 days a week for 12 months.
  Interventions: Behavioral: physical exercise programme
- Standard of care (No Intervention): They will have all the follow-up provided by the hospital in the same way as the intervention group in addition to the relevant assessments carried out throughout the clinical trial, throughout the study they will be encouraged to have an active lifestyle.

INTERVENTIONS:
Behavioral: physical exercise programme — patients undergoing bariatric surgery who have undergone a post-operative supervised physical exercise programme and no exercise programme.
  Arms: physical exercise program

SUMMARY:
CLINICAL TRIAL ON THE EFFECT OF SUPERVISED PHYSICAL EXERCISE AFTER BARIATRIC SURGERY ON MUSCLE MASS AND BONE DENSITY (OBEFIT STUDY)

DETAILED DESCRIPTION:
Introduction Background and rationale Obesity is currently a complex disease that has reached pandemic proportions and affects millions of people worldwide. Bariatric surgery can generate adverse side effects such as loss of bone mineral density, loss of muscle mass, reduction in cardiorespiratory capacity. Therefore, accompanying medical treatment with an individualised physical exercise intervention can generate a multitude of health benefits for the patient.

Objectives

As main objective the investigators focus on:

- To determine the differences in muscle mass and bone density in patients undergoing bariatric surgery who have undergone a post-operative supervised physical exercise programme and no exercise programme.

* To determine the differences in muscle function using the hand grip test.
* To determine BMD loss using densitometry.

Secondary objectives:

* To analyse maximal fat oxidation throughout the whole process from metabolic inflexibility to metabolic flexibility).
* To determine differences in body composition.
* To determine the resolution of type 2 diabetes mellitus and arterial hypertension (AHT).
* To determine the improvement in quality of life by means of an accredited test.

Null hypothesis:

1. There are no differences in muscle mass and bone density in patients who undergo supervised physical exercise postoperatively versus patients who do not exercise.

Alternative hypothesis:

1. There are differences in muscle mass and bone density in patients undergoing supervised physical exercise postoperatively versus non-exercising patients.

Trial design The trial will consist of a randomised controlled study of patients currently on the surgical waiting list for bariatric surgery who meet the inclusion criteria until the sample size is completed.

Two groups (control and intervention) will be established and will come in waves.

Methods Participants, interventions and results Scope of the study The assessment and intervention of the study will take place at the Pablo de Olavide University in Seville. The medical assessment and surgical intervention will be carried out at the General and Digestive System Surgery Management Unit of the Virgen del Rocío University Hospital in Seville.

ELIGIBILITY:
INCLUSION CRITERIA

Patients who are on the waiting list for bariatric surgery (gastric bypass or sleeve) at the Hospital Universitario Virgen del Rocío in Seville, in addition to:

* Be 18 years of age or older.
* Suitable for physical exercise.
* Signature of informed consent. EXCLUSION CRITERIA.
* Body weight greater than 150kg.
* Distance from the place of residence to the Pablo de Olavide University in Seville greater than 60 km or 45 minutes by car.
* Having any of the following conditions: lipedema, cancer survivors, metabolic bone diseases, consumption of medication or presence of pathology that affects bone health.
* Patients undergoing dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Differences in muscle mass | 12 months
  To determine the differences in muscle mass and bone density in patients undergoing bariatric surgery who have undergone a post-operative supervised physical exercise programme and no exercise programme.
  o To determine the differences in muscle function using the hand grip test.

OTHER OUTCOMES:
differences in bone density | 12 months
  To determine the differences in bone density in patients undergoing bariatric surgery who have undergone a post-operative supervised physical exercise programme and no exercise programme.
  o To determine BMD loss using densitometry.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital virgen del rocio, Seville, Sevilla
  - Universidad Pablo de Olavide, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: Undecided